CLINICAL TRIAL: NCT00279266
Title: A Randomized Double Blinded Pilot Study of Oral Thiamine in the Symptomatic Treatment of Painful Diabetic Peripheral Neuropathy
Brief Title: Oral Thiamine for the Treatment of Painful Diabetic Peripheral Neuropathy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: inadequate recruitment
Sponsor: Loma Linda University (Other)
Responsible Party: Principal Investigator, Travis Losey, Assistant Professor of Neurology, Loma Linda University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 55288
Record Dates: First submitted 2006-01-18; First posted 2006-01-19 (Estimated); Last update posted 2015-05-13 (Estimated); Status verified 2015-05

CONDITIONS: Peripheral Neuropathy; Diabetes Mellitus; Diabetes Complications
Keywords: Diabetic Peripheral Neuropathy; Peripheral Neuropathy; Diabetes Mellitus
MeSH Terms: conditions — Peripheral Nervous System Diseases; Diabetes Mellitus; Diabetes Complications | interventions — Thiamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Thiamine

SUMMARY:
This study will examine the effect of oral thiamine (Vitamin B1) supplementation on pain in patients with diabetic peripheral neuropathy.

DETAILED DESCRIPTION:
It is estimated that more then 5 million people in the United States suffer from Diabetes Mellitus, and of these up to 80% suffer from painful diabetic peripheral neuropathy. Multiple medications have been tried for the treatment of painful diabetic neuropathy. These medications are directed at symptomatic relief and do not address the underlying cause of painful peripheral neuropathy. Thiamine is a water-soluble vitamin that participates in carbohydrate metabolism. Deficiency of thiamine causes beriberi, characterized by painful peripheral neuropathy and cardiomyopathy. Basic research has suggested that thiamine deficiency may also be involved in the etiology of diabetic neuropathy by preventing the glycation of nerve fibers as well as apoptosis of endothelial cells. A study in the developing world found that oral thiamine and pyridoxine were helpful in improving the pain experienced in diabetic peripheral neuropathy as well as improving signs of neuropathy seen on neurological examination. A screening study of patients with type II diabetes found that 76% of patients tested had a low serum thiamine level.

Our study will examine the effect of oral thiamine supplementation on the symptom of pain in painful diabetic peripheral neuropathy. In addition we will follow serum thiamine levels to see if clinical change correlates with changes in serum thiamine levels

ELIGIBILITY:
Inclusion Criteria:

Diagnosis of Diabetes Mellitus Painful diabetic neuropathy for > six months with a score of >40mm on a visual pain analog scale Age >18 years Hemoglobin A1c obtained within the last 3 months. Willingness and ability to comply with the study requirements and give informed consent.

Exclusion Criteria:

Known history of alcohol abuse, recreational drug abuse, thyroid dysfunction, syphilis, multiple myeloma, known nutrient deficiency, history of gastric bypass surgery or HIV. Hgb A1c>11

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-01; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Daily pain evaluations on a visual analog pain scale

SECONDARY OUTCOMES:
Pain over the last 7 days as recorded on a Visual Analog pain scale
Changes in Sf-36v2 results
Changes in blood thiamine levels
Changes in the McGill short form pain questionnaire
Changes in sleep disturbance in secondary to pain as rated by a visual analog scale

CONTACTS AND LOCATIONS:
Overall Officials: Rodolfo Escutin, MD, Principal Investigator — Loma Linda University
Locations (1):
- Loma Linda University Department of Neurology, Loma Linda, California, United States

REFERENCES:
- [Background] Thornalley PJ. Glycation in diabetic neuropathy: characteristics, consequences, causes, and therapeutic options. Int Rev Neurobiol. 2002;50:37-57. doi: 10.1016/s0074-7742(02)50072-6. PMID 12198817
- [Background] Abbas ZG, Swai AB. Evaluation of the efficacy of thiamine and pyridoxine in the treatment of symptomatic diabetic peripheral neuropathy. East Afr Med J. 1997 Dec;74(12):803-8. PMID 9557427